CLINICAL TRIAL: NCT00929643
Title: The Impact Of Bacterial Resistance On Healthcare Costs For Hospitalized Patients With Complicated Intra-Abdominal Infections
Brief Title: Impact Of Bacterial Resistance On Healthcare Costs For Hospitalized Patients With Complicated Intra-Abdominal Infections
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3074A1-102311; B1811060
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Results first posted 2012-08-06 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Complicated Intra-Abdominal Infection
Keywords: health care costs; Intra-Abdominal Infection
MeSH Terms: conditions — Intraabdominal Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — success of the initial empiric treatment

SUMMARY:
The objective of this study is to estimate the costs of empiric antibiotic therapy and hospitalization costs for patients with a complicated intra-abdominal infection, and to assess the impact of treatment failure of initial antibiotic empiric therapy on pharmacological and total healthcare costs for these patients in Greece.

DETAILED DESCRIPTION:
Every patient diagnosed with complicated intra-abdominal infections will enter the study, until the pre-specified number of patients is reached. Patients diagnosed with any of conditions mentioned below (inclusion criteria) will enter the study, until the pre-specified number of patients is reached.

ELIGIBILITY:
Inclusion Criteria:

* A recorded primary diagnosis of a complicated intra-abdominal. infection (cIAI) and a procedure involving a laparotomy, laparoscopy, or percutaneous drainage of an intra-abdominal abscess The study will be a prospective, multi-centre, epidemiological study of patients (aged > 18 years) diagnosed with a complicated intra-abdominal infection AND who received a procedure involving laparotomy/laparoscopy or percutaneous drainage of an intra-abdominal abscess. cIAI's will include the following conditions/ diagnoses:
* Gastric ulcer with perforation;
* Gastric ulcer with hemorrhage and perforation;
* Duodenal ulcer with perforation;
* Duodenal ulcer with hemorrhage and perforation;
* Peptic ulcer with perforation;
* Peptic ulcer with hemorrhage and perforation;
* Gastrojejunal ulcer with perforation;
* Gastrojejunal ulcer with hemorrhage and perforation;
* Acute appendicitis with generalized peritonitis;
* Acute appendicitis with peritoneal abscess;
* Peritonitis;
* Abscess of intestine;
* Fistula of intestine, excluding rectum and anus;
* Ulceration of intestine;
* Perforation of intestine;
* Abscess of liver; or
* Acute cholecystitis with perforation.

The initial antibiotic regimen will be defined as all IV antibiotics newly received either on the day immediately prior to laparotomy or laparoscopy or percutaneous drainage of an intra-abdominal abscess, or on the day of these procedures, given that the use of these procedures prior to initiation of IV antibiotic regimens in complicated IAIs , which is increasingly common, is likely reflective of prophylaxis.

Exclusion Criteria:

* Patients not signing an informed consent form.
* Patients participating in another interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for complicated intra-abdominal infections
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Greece (9):
  - Pfizer Investigational Site, Athens, Athens
  - Pfizer Investigational Site, Cholargós, Athens
  - Pfizer Investigational Site, Haidari, Athens
  - Pfizer Investigational Site, Marousi, Athens
  - Pfizer Investigational Site, N. Ionia, Athens
  - Pfizer Investigational Site, Peireus, Athens
  - Pfizer Investigational Site, Rio, Patras
  - Pfizer Investigational Site, Thessaloniki, Thessaloniki
  - Pfizer Investigational Site, Heraklion, Vrete

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3074A1-102311&StudyName=Impact%20Of%20Bacterial%20Resistance%20On%20Healthcare%20Costs%20For%20Hospitalized%20Patients%20With%20Complicated%20Intra-Abdominal%20Infections

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Observational, epidemiological, noninterventional study.
Groups:
- All Enrolled Participants: Hospitalized participants over 18 years of age, diagnosed with complicated intra-abdominal infections (cIAIs) who had received a procedure involving laparotomy/laparoscopy or percutaneous drainage of an intra-abdominal abscess; treatment followed standard clinical practice.
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 203
Completed | 201
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 201
Age Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 136

OUTCOME MEASURES:

1. Primary Outcome: Duration of Hospitalization
Description: Overall health care resource utilization was analyzed using mean duration of hospitalization.
Time Frame: Baseline up to 6 months
Population: Full Analysis Set (FAS): All enrolled participants who fulfilled the protocol inclusion criteria. N=number of participants with nonmissing data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 193
Days | 14.1 (12.7)

2. Primary Outcome: Percentage of Participants With Initial Empiric Antibiotic Therapy (by Therapeutic Class)
Time Frame: Baseline up to 6 months
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 201
Percentage of participants
  Metronidazole | 59.2
  b-Lactamase Inhibitors (BLI) | 38.3
  Cephalosporines (2nd generation) | 30.3
  Quinolones | 16.9
  Aminoglycocides | 12.4
  Carbapenems | 8.5
  Glycopeptides | 8.0
  Glycycyclines | 5.0
  Antifungals | 4.0
  Cephalosporines (3rd generation) | 4.0
  Lipopeptides/oxazolidinones | 2.0
  Clindamycin | 1.5
  Beta lactams | 0.5
  Cephalosporines (4th generation) | 0.5
  Other | 0.5

3. Primary Outcome: Percentage of Participants With Failure of Initial Empiric Antibiotic Therapy
Description: Failure of initial empiric therapy was assessed by an independent committee of qualified healthcare professionals (surgeon, and microbiologist specialist) and defined as requirement of additional antibiotic or change in antibacterial therapy on any day following the initial laparotomy, laparoscopy, or percutaneous drainage; or additional laparotomy, laparoscopy, or percutaneous drainage at least 2 days following the initial surgical/radiological intervention; or participant death due to infection.
Time Frame: Baseline up to 6 months
Population: FAS; n=number of participants in which failure could be assessed
Measure: Number; unit: Percentage of participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 196
Percentage of participants | 42.9

4. Primary Outcome: Duration of Hospitalization (by Failure of Initial Empiric Treatment)
Description: Yes equals (=) initial empiric antibiotic treatment failed (additional antibiotic therapy or a change in antibacterial therapy was required following laparotomy/laparoscopy or percutaneous draininge or participant died due to infection); No=initial empiric antibiotic treatment successful (infectious process resolved and no change in initial empiric antibiotic therapy was required during the course of hospitalization except for stepdown therapy, de-escalation or intravenous to oral switch).
Time Frame: Baseline up to 6 months
Population: FAS; n=number of participants with nonmissing data
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 189
Days
  No (n=111) | 8.9 (4.5)
  Yes (n=78) | 21.9 (16.4)

5. Secondary Outcome: Percentage of Participants With Specific Pathogen
Time Frame: Baseline up to 6 months
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 201
Percentage of participants
  Escherichia coli | 23.9
  Pseudomonas aeruginosa | 9.5
  Klebsiella pneumoniae | 9.0
  Acinetobacter baumanii | 8.5
  Staphylococcus (S.) aureus (methicillin sensitive) | 1.5
  S. aureus (methicillin resistant) | 1.0
  Stenotrophomonas | 0.5
  Candida albicans | 7.5
  Candida species (spp) (non Albicans) | 1.5
  Fungi without species identification | 0.5
  S. epidermis | 2.5
  S. hominis | 2.5
  S. haemolyticus | 1.0
  S. lentus | 0.5
  S. intermedius | 0.5
  Enterococcus faecalis | 10.9
  Enterococcus faecium | 7.0
  Enterococcus durans | 0.5
  Enterococcus spp (vancomycin resistant) | 2.0
  Streptococcus viridans | 1.5
  Streptococcus salivarius | 1.0
  Streptococcus haemolyticus | 1.0
  Streptococcus mitis | 1.0
  Streptococcus pneumoniae | 0.5
  Streptococcus pyogenes | 0.5
  Streptococcus group C | 0.5
  Streptococcus Bovis | 0.5
  Streptococcus acidominimus | 0.5
  Bacteroides fragilis group | 4.0
  Enterobacter spp | 2.0
  Proteus spp | 2.0
  Proteus mirabilis | 2.0
  Bacteroides spp. (non fragilis) | 1.0
  Aeromonas hydrophila | 1.0
  Hafnia alvei | 1.0
  Enterobacter cloacae | 1.0
  Citrobacter braakii | 1.0
  Haemophilus spp | 0.5
  Morganella morganii | 0.5
  Prevotella bivia | 0.5
  Peptostreptococcus | 0.5
  Prevotella intermedia | 0.5
  Prevotella oralis | 0.5
  Actinomyces israelii | 0.5
  Enterobacter aerogenes | 0.5
  Ralstonia mannitolilytica | 0.5
  Comamonas acidovorans | 0.5
  Comamonas spp | 0.5
  Prevotella species | 0.5
  Citrobacter freundii | 0.5

6. Secondary Outcome: Percentage of Participants by Diagnosis at Discharge
Time Frame: Month 6 or study exit
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 201
Percentage of participants
  Perforation of intestine | 15.9
  Acute appendicitis with (w/) peritoneal abscess | 13.4
  Postoperative peritonitis | 13.4
  Acute cholecystitis w/perforation | 10.4
  Acute appendicitis w/generalized peritionitis | 10.0
  Gastric ulcer w/ perforation | 9.5
  Duodenal ulcer w/perforation | 7.0
  Abscess of liver | 4.5
  Diverticulitis complicated | 4.5
  Fistula of intestine, excluding rectum and anus | 3.0
  cIAI: abdominal neplasm surgical extract/decrease | 3.0
  Gastrojejunal ulcer w/perforation | 2.5
  Gastrojejunal ulcer w/hemorrhage and perforatio | 2.0
  Abscess of intestine | 2.0
  Gastric ulcer w/hemorrhage and perforation | 1.0
  Peptic ulcer w/perforation | 0.5
  Peritonitis | 0.5
  Other | 8.0

ADVERSE EVENTS:
Description: Adverse event (AE) data were collected retrospectively by reviewing medical records using data available until December 2010. All death reports were sent to the Sponsor as case report forms upon identification in the database. In addition, the investigator retrospectively completed an AE/serious adverse event (SAE) form for any suspected AEs/SAEs.
Arm/Group | All Enrolled Participants
Serious Adverse Events (participants affected / at risk) | 20/201
Other Adverse Events (participants affected / at risk) | 0/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Enrolled Participants (N=201)
Unknown cause of death (General disorders) | 6
Multi-organ failure (General disorders) | 5
Systemic inflammatory response syndrome (General disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 2
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Subdiaphragmatic abscess (Gastrointestinal disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiorespiratory arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Cardiorespiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Gallbladder perforation (Hepatobiliary disorders) | 1
Anastomotic complication (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.